CLINICAL TRIAL: NCT04144270
Title: The Importance of Muscle Function in Patients With Disseminated Bladder Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Roche Pharma AG (Industry); Merck Sharp & Dohme LLC (Industry); Beckett Foundation (Other); Onkologisk Forskningsfond (Unknown)
Responsible Party: Principal Investigator, Lise Hoej Omland, MD, Rigshospitalet, Denmark
Other Study IDs: 70298
Record Dates: First submitted 2019-10-01; First posted 2019-10-30 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Urinary Bladder Neoplasm
Keywords: Urinary Bladder Neoplasm; Urothelium Neoplasm; Oncology; Muscle function; Sarcopenia
MeSH Terms: conditions — Urinary Bladder Neoplasms; Neoplasms; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Included patients: One-arm study. All included patients will have muscle mass and muscle function evaluated
  Interventions: Other: Evaluation of muscle mass and muscle function

INTERVENTIONS:
Other: Evaluation of muscle mass and muscle function — Included patients have their muscle mass and muscle function evaluated before start on and after completion of oncological treatment.

SUMMARY:
This study investigates if reduced muscle mass and muscle function predispose to poor completion of oncological treatment in patients with bladder cancer (including cancer of the renal pelvis, ureter and urethra) and if muscle mass and muscle function change during oncological treatment in these patients. It also evaluates biomarkers for sarcopenia.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age ≥ 18 år
* Histologically verified cancer of the renal pelvis, ureter, bladder or urethra regardless of type of histology
* ECOG performance status 0 - 3
* Meet the requirements for receiving oncological treatment (neoadjuvant chemotherapy for localized disease, chemotherapy or immunotherapy for disseminated disease).

Exclusion Criteria:

* Age < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with localized cancer in the urinary tract undergoing neoadjuvant chemotherapy prior to radical cystektomy or patients with disseminated disease undergoing chemotherapy or immunotherapy. Patients are identified and included from Department of Oncology, Rigshospitalet, Copenhagen, Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-11-18 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Muscle mass | Up to 36 months
  We will describe if muscle mass at baseline is correlated to completion of planned systemic oncological treatment

SECONDARY OUTCOMES:
Muscle strength | Up to 36 months
  We will describe if muscle strength at baseline is correlated to completion of planned systemic oncological treatment
Muscle mass changes during systemic oncological treatment | Up to 36 months
  We will describe if muscle mass change during systemic oncological treatment
Muscle strength changes during systemic oncological treatment | Up to 36 months
  We will describe if muscle mass change during systemic oncological treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lise Hoej Omland, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No